CLINICAL TRIAL: NCT05861687
Title: Comparative Recurrence Rate Investigation of Esomeprazole Versus Lansoprazole in Triple-Combination Therapy to Eradicate Helicobacter Pylori Infection Among Pediatrics: Multicentre, Randomized, and Controlled Trials
Brief Title: Recurrence Rate Comparison Between Esomeprazole and Lansoprazole in Eradicating Helicobacter Pylori Infection Among Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Finni Kollins (Other)
Responsible Party: Sponsor-Investigator, Finni Kollins, Resident Doctor, Universitas Sumatera Utara
Organization: Universitas Sumatera Utara (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LB.02.01.XV.III.2.2.2/344/2022
Record Dates: First submitted 2023-05-06; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Triple therapy; Children; Esomeprazole; Lansoprazole
MeSH Terms: interventions — Esomeprazole; Lansoprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esomeprazole in combination with Amoxicillin and Clarithromycin (Experimental): Esomeprazole : once a day per oral; 0.4 mg/kg Amoxicillin: thrice a day per oral; 25 mg/kg Clarithromycin: twice a day per-oral; 7.5 mg/kg
  Interventions: Drug: Esomeprazole; Drug: Amoxicillin; Drug: Clarithromycin
- Lansoprazole in combination with Amoxicillin and Clarithromycin (Active Comparator): Lansoprazole: once a day per oral; 15 mg if body weight < 30 kg and 30 mg if body weight > 30 kg Amoxicillin: thrice a day per oral; 25 mg/kg Clarithromycin: twice a day per-oral; 7.5 mg/kg
  Interventions: Drug: Lansoprazole; Drug: Amoxicillin; Drug: Clarithromycin

INTERVENTIONS:
Drug: Esomeprazole — Administered once a day per-oral (PO) with the dose of 0.4 mg/kg
  Arms: Esomeprazole in combination with Amoxicillin and Clarithromycin
Drug: Lansoprazole — Administered once a day per-oral (PO) with the dose of 15 mg if individual's body mass was <30 kg, and 30 mg if it was >30 kg
  Arms: Lansoprazole in combination with Amoxicillin and Clarithromycin
Drug: Amoxicillin — Administered thrice a day per-oral (PO) with the dose of 25 mg/kg
Drug: Clarithromycin — Administered twice a day per-oral with the dose of 7.5 mg/kg

SUMMARY:
This study aims to compare the recurrence rates of Esomeprazole and Lansoprazole in triple combination therapy to eradicate H.pylori infection in children. The participants were divided into two groups, those who received Esomeprazole and those who received Lansoprazole

DETAILED DESCRIPTION:
H. pylori eradication therapy is still contentious. A treatment that is uncomplicated, well-tolerated, and boasts an efficiency rate of more than 80% is recommended.

PPIs are a type of acid-sensitive drug which is most beneficial in preventing the degradation of drugs in the stomach. In developing countries, Esomeprazole and Lansoprazole were mainly selected as a drug of choice. Major influential factors such as Esomeprazole's additional antioxidant ability, are comparable to vitamin C. This is due to its ability to scavenge Diphenyl Picrylhydrazyl (DPPH) free radicals at low concentrations. Lansoprazole also possess similar ability, albeit needs a slightly higher concentration to reach a similar effect. In terms of IC50 values, both drugs have a substantial advantage over vitamin C, earning them the title of 'potentially ideal' agents in the treatment algorithm. Furthermore, numerous studies mention that children better tolerate PPIs.

ELIGIBILITY:
Inclusion Criteria:

* Subject has positive clinical symptoms (gastrointestinal pain, nausea, vomiting, hematemesis, or melena)
* Subject had been diagnosed with H.pylori infection prior to endoscopy and rapid urease testing

Exclusion Criteria:

* subject has a history of using antibiotics or non-steroidal anti-inflammatory medicines (NSAIDs) within 14 days prior to surgery
* subject has a concomitant systemic disease (e.g., renal failure, liver cirrhosis, cancer, etc.) that could theoretically affect the subject's response to treatment
* Incomplete triple pharmacologic treatment due to the subject's lack of medication adherence

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori Stool Antigen Test | 15 days
  The stool of the subjects will be assessed on day-15 after drug administration. A negative result indicates that patient is infection-free

SECONDARY OUTCOMES:
Helicobacter pylori Stool Antigen Test | 75 days
  The stool of the subjects will be analyzed on day-90 after drug administration to assess whether a reinfection is present. A negative result indicates that patient is infection-free

CONTACTS AND LOCATIONS:
Locations (2):
- Indonesia (2):
  - Universitas Sumatera Utara General Hospital, Medan, North Sumatera
  - Haji Adam Malik General Hospital, Medan, North Sumatera

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awuku YA, Simpong DL, Alhassan IK, Tuoyire DA, Afaa T, Adu P. Prevalence of helicobacter pylori infection among children living in a rural setting in Sub-Saharan Africa. BMC Public Health. 2017 Apr 24;17(1):360. doi: 10.1186/s12889-017-4274-z. PMID 28438158
- [Background] Jafar S, Jalil A, Soheila N, Sirous S. Prevalence of helicobacter pylori infection in children, a population-based cross-sectional study in west iran. Iran J Pediatr. 2013 Feb;23(1):13-8. PMID 23550042
- [Background] Allen SJ, Thomas JE, Alexander ND, Bailey R, Emerson PM. Flies and Helicobacter pylori infection. Arch Dis Child. 2004 Nov;89(11):1037-8. doi: 10.1136/adc.2003.045880. PMID 15499059
- [Background] Mansour MM, Al Hadidi KhM, Omar MA. Helicobacter pylori and recurrent abdominal pain in children: is there any relation? Trop Gastroenterol. 2012 Jan-Mar;33(1):55-61. doi: 10.7869/tg.2012.9. PMID 22803297
- [Background] Das BK, Kakkar S, Dixit VK, Kumar M, Nath G, Mishra OP. Helicobacter pylori infection and recurrent abdominal pain in children. J Trop Pediatr. 2003 Aug;49(4):250-2. doi: 10.1093/tropej/49.4.250. PMID 12929890
- [Background] Quek SH. Recurrent abdominal pain in children: a clinical approach. Singapore Med J. 2015 Mar;56(3):125-8; quiz 132. doi: 10.11622/smedj.2015038. PMID 25820843
- [Background] Jones NL, Koletzko S, Goodman K, Bontems P, Cadranel S, Casswall T, Czinn S, Gold BD, Guarner J, Elitsur Y, Homan M, Kalach N, Kori M, Madrazo A, Megraud F, Papadopoulou A, Rowland M; ESPGHAN, NASPGHAN. Joint ESPGHAN/NASPGHAN Guidelines for the Management of Helicobacter pylori in Children and Adolescents (Update 2016). J Pediatr Gastroenterol Nutr. 2017 Jun;64(6):991-1003. doi: 10.1097/MPG.0000000000001594. PMID 28541262
- [Background] Urgesi R, Cianci R, Riccioni ME. Update on triple therapy for eradication of Helicobacter pylori: current status of the art. Clin Exp Gastroenterol. 2012;5:151-7. doi: 10.2147/CEG.S25416. Epub 2012 Sep 17. PMID 23028235
- [Background] Sahara S, Sugimoto M, Uotani T, Ichikawa H, Yamade M, Iwaizumi M, Yamada T, Osawa S, Sugimoto K, Umemura K, Miyajima H, Furuta T. Twice-daily dosing of esomeprazole effectively inhibits acid secretion in CYP2C19 rapid metabolisers compared with twice-daily omeprazole, rabeprazole or lansoprazole. Aliment Pharmacol Ther. 2013 Nov;38(9):1129-37. doi: 10.1111/apt.12492. Epub 2013 Sep 16. PMID 24099474
- [Background] Peterson WL. The role of antisecretory drugs in the treatment of Helicobacter pylori infection. Aliment Pharmacol Ther. 1997 Apr;11 Suppl 1:21-5. doi: 10.1046/j.1365-2036.11.s1.4.x. PMID 9146787
- [Background] Ward RM, Kearns GL. Proton pump inhibitors in pediatrics : mechanism of action, pharmacokinetics, pharmacogenetics, and pharmacodynamics. Paediatr Drugs. 2013 Apr;15(2):119-31. doi: 10.1007/s40272-013-0012-x. PMID 23512128
- [Background] Nishida T, Tsujii M, Tanimura H, Tsutsui S, Tsuji S, Takeda A, Inoue A, Fukui H, Yoshio T, Kishida O, Ogawa H, Oshita M, Kobayashi I, Zushi S, Ichiba M, Uenoyama N, Yasunaga Y, Ishihara R, Yura M, Komori M, Egawa S, Iijima H, Takehara T. Comparative study of esomeprazole and lansoprazole in triple therapy for eradication of Helicobacter pylori in Japan. World J Gastroenterol. 2014 Apr 21;20(15):4362-9. doi: 10.3748/wjg.v20.i15.4362. PMID 24764674
- [Background] Niv Y. H pylori recurrence after successful eradication. World J Gastroenterol. 2008 Mar 14;14(10):1477-8. doi: 10.3748/wjg.14.1477. PMID 18330934
- [Background] Halitim F, Vincent P, Michaud L, Kalach N, Guimber D, Boman F, Turck D, Gottrand F. High rate of Helicobacter pylori reinfection in children and adolescents. Helicobacter. 2006 Jun;11(3):168-72. doi: 10.1111/j.1523-5378.2006.00396.x. PMID 16684264
- [Background] Ding Z, Zhao S, Gong S, Li Z, Mao M, Xu X, Zhou L. Prevalence and risk factors of Helicobacter pylori infection in asymptomatic Chinese children: a prospective, cross-sectional, population-based study. Aliment Pharmacol Ther. 2015 Oct;42(8):1019-26. doi: 10.1111/apt.13364. Epub 2015 Aug 14. PMID 26271484
- [Background] Leal-Herrera Y, Torres J, Monath TP, Ramos I, Gomez A, Madrazo-de la Garza A, Dehesa-Violante M, Munoz O. High rates of recurrence and of transient reinfections of Helicobacter pylori in a population with high prevalence of infection. Am J Gastroenterol. 2003 Nov;98(11):2395-402. doi: 10.1111/j.1572-0241.2003.07708.x. PMID 14638339
- [Background] Sheu BS, Kao AW, Cheng HC, Hunag SF, Chen TW, Lu CC, Wu JJ. Esomeprazole 40 mg twice daily in triple therapy and the efficacy of Helicobacter pylori eradication related to CYP2C19 metabolism. Aliment Pharmacol Ther. 2005 Feb 1;21(3):283-8. doi: 10.1111/j.1365-2036.2005.02281.x. PMID 15691303
- [Background] Kawabata H, Habu Y, Tomioka H, Kutsumi H, Kobayashi M, Oyasu K, Hayakumo T, Mizuno S, Kiyota K, Nakajima M, Kimoto K, Inokuchi H, Kawai K. Effect of different proton pump inhibitors, differences in CYP2C19 genotype and antibiotic resistance on the eradication rate of Helicobacter pylori infection by a 1-week regimen of proton pump inhibitor, amoxicillin and clarithromycin. Aliment Pharmacol Ther. 2003 Jan;17(2):259-64. doi: 10.1046/j.1365-2036.2003.01406.x. PMID 12534411
- [Background] Mainz D, Borner K, Koeppe P, Kotwas J, Lode H. Pharmacokinetics of lansoprazole, amoxicillin and clarithromycin after simultaneous and single administration. J Antimicrob Chemother. 2002 Nov;50(5):699-706. doi: 10.1093/jac/dkf172. PMID 12407126
- [Background] Liou JM, Chen CC, Chang CM, Fang YJ, Bair MJ, Chen PY, Chang CY, Hsu YC, Chen MJ, Chen CC, Lee JY, Yang TH, Luo JC, Chen CY, Hsu WF, Chen YN, Wu JY, Lin JT, Lu TP, Chuang EY, El-Omar EM, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Long-term changes of gut microbiota, antibiotic resistance, and metabolic parameters after Helicobacter pylori eradication: a multicentre, open-label, randomised trial. Lancet Infect Dis. 2019 Oct;19(10):1109-1120. doi: 10.1016/S1473-3099(19)30272-5. PMID 31559966
- [Background] Perez-Cobas AE, Gosalbes MJ, Friedrichs A, Knecht H, Artacho A, Eismann K, Otto W, Rojo D, Bargiela R, von Bergen M, Neulinger SC, Daumer C, Heinsen FA, Latorre A, Barbas C, Seifert J, dos Santos VM, Ott SJ, Ferrer M, Moya A. Gut microbiota disturbance during antibiotic therapy: a multi-omic approach. Gut. 2013 Nov;62(11):1591-601. doi: 10.1136/gutjnl-2012-303184. Epub 2012 Dec 12. PMID 23236009
- [Background] Katsuki H, Nakamura C, Arimori K, Fujiyama S, Nakano M. Genetic polymorphism of CYP2C19 and lansoprazole pharmacokinetics in Japanese subjects. Eur J Clin Pharmacol. 1997;52(5):391-6. doi: 10.1007/s002280050307. PMID 9272410
- [Background] Wu L, Wang Z, Sun G, Peng L, Lu Z, Yan B, Huang K, Yang Y. Effects of anti-H. pylori triple therapy and a probiotic complex on intestinal microbiota in duodenal ulcer. Sci Rep. 2019 Sep 6;9(1):12874. doi: 10.1038/s41598-019-49415-3. PMID 31492912
- [Background] Park SK, Park DI, Choi JS, Kang MS, Park JH, Kim HJ, Cho YK, Sohn CI, Jeon WK, Kim BI. The effect of probiotics on Helicobacter pylori eradication. Hepatogastroenterology. 2007 Oct-Nov;54(79):2032-6. PMID 18251154
- [Background] Dai C, Zheng CQ, Jiang M. Efficacy of probiotics in Helicobacter pylori eradication therapy. J Clin Gastroenterol. 2013 Oct;47(9):814-5. doi: 10.1097/MCG.0b013e318298a32c. No abstract available. PMID 23751838
- [Background] Lynch SV, Pedersen O. The Human Intestinal Microbiome in Health and Disease. N Engl J Med. 2016 Dec 15;375(24):2369-2379. doi: 10.1056/NEJMra1600266. No abstract available. PMID 27974040
- [Background] Gisbert JP, Pajares JM. Stool antigen test for the diagnosis of Helicobacter pylori infection: a systematic review. Helicobacter. 2004 Aug;9(4):347-68. doi: 10.1111/j.1083-4389.2004.00235.x. PMID 15270750
- [Background] Vaira D, Malfertheiner P, Megraud F, Axon AT, Deltenre M, Hirschl AM, Gasbarrini G, O'Morain C, Garcia JM, Quina M, Tytgat GN. Diagnosis of Helicobacter pylori infection with a new non-invasive antigen-based assay. HpSA European study group. Lancet. 1999 Jul 3;354(9172):30-3. doi: 10.1016/s0140-6736(98)08103-3. PMID 10406362
- [Background] Yang HR. Updates on the Diagnosis of Helicobacter pylori Infection in Children: What Are the Differences between Adults and Children? Pediatr Gastroenterol Hepatol Nutr. 2016 Jun;19(2):96-103. doi: 10.5223/pghn.2016.19.2.96. Epub 2016 Jun 28. PMID 27437185